CLINICAL TRIAL: NCT03116243
Title: Migrant and Seasonal Head Start (MSHS) Study
Brief Title: Migrant and Seasonal Head Start Study
Acronym: MSHS
Status: Completed | Type: Observational
Sponsor: Abt Associates (Industry)
Collaborators: The Catholic University of America (Other); Westat (Other)
Responsible Party: Sponsor
Other Study IDs: MSHS
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2017-04

CONDITIONS: Migrant and Seasonal Head Start
Keywords: migrant and seasonal head start; early childhood education; head start

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MSHS children and families: Cohort includes:
  * children (1272)
  * parents (1272)
  * teachers (159)
  * teaching assistants (159)
  * program and center directors (253)

SUMMARY:
The MSHS Study is a nationally representative study commissioned by the U.S. Office of Health and Human Services' Administration for Children and Families that will describe the characteristics and experiences of the children and families who enroll in MSHS and the practices and services of the MSHS programs that serve them. The MSHS Study draws heavily on the Design for MSHS Survey Report (2011) and is informed by the current context of key policy and programmatic issues and broader issues impacting the lives of migrant and seasonal farmworkers and their families.

The MSHS Study has two components: a Program/Center component and a Classroom, Family, Child component that are based on distinct samples. The first component is off-site and consists of mailed surveys that will be sent to the universe of MSHS program directors and a representative subset of center directors to provide information on program and center operations. The second component consists of onsite data collection - including classroom observations, surveys with teachers and assistant teachers, parent interviews, teacher and parent child reports, and direct child assessments - with a nationally-representative sample of centers, classrooms, families and children.

Once data are collected, the study will address a set of research questions that can be summarized into three broad categories: (1) What are the characteristics of MSHS programs, families, and children? (2) What services do MSHS programs provide, what instructional and language practices are used, and what is the quality of MSHS classrooms? and (3) What are the associations between MSHS characteristics and child/family well-being?

ELIGIBILITY:
Inclusion Criteria:

* infants, toddlers, and preschoolers in participating Migrant and Seasonal Head Start centers/classrooms across the U.S. and their teachers and parents. Also includes center directors and program directors.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes children birth to five years who attend Migrant Seasonal Head Start (MSHS) programs, along with their parents and teachers, center directors, and program directors.
Sampling Method: Probability Sample
Enrollment: 1404 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Language Literacy | 1 year
  Indicators of language literacy will be assessed during week-long site visits using Letter-Word Identification & "Identificación de letras y palabras" in the Woodcock-Muñoz Language Survey.
Emergent Literacy | 1 year
  Indicators of emergent literacy will be assessed during week-long site visits using the Spanish Version (or English version for children who are not Spanish speakers) of the PLS-5 Auditory Comprehension subscale.
Emotional Skills | 1 year
  Indicators of emotional skills will be assessed during week-long site visits using the Cognitive/ Social and Emotional/Regulations Scales from the Leiter-Third Edition Examiner Rating Scales.
Classroom Quality | 1 year
  Classroom quality will be assessed during the week-long site visits using the Early Language and Literacy Classroom Observation (ELLCO) Tool and the Classroom Assessment Scoring System™ (CLASS™).

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Barrueco, Ph.D., Principal Investigator — The Catholic Univeristy of America; Michael L Lopez, Ph.D., Principal Investigator — Abt Associates; Linda Caswell, Ed.D., Study Director — Abt Associates
Locations (1):
- Abt Associates, Inc., Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
The MSHS Study team will prepare restricted use datasets and documentation, to be archived with a data storage site such as the Inter-university Consortium for Political and Social Research (ICPSR) at the University of Michigan, so that future researchers may use the MSHS Study data to replicate findings and explore new areas of inquiry.

REFERENCES:
- [Background] O'Brien RW, Barrueco S, Lopez ML, D'Elio ML. Design for Migrant and Seasonal Head Start Survey. Washington, D.C.: Administration for Children and Families, 2011.